CLINICAL TRIAL: NCT01514682
Title: Anti-Inflammatory Combination Therapy for the Treatment of Schizophrenia
Brief Title: Anti-Inflammatory Treatment of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00051603; 11T-002
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; anti-inflammatory; salsalate; statins; omega-3-fatty acids
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo pills to be assigned using a permuted randomization system
  Interventions: Drug: Placebo
- Anti-inflammatory Combination Therapy (Experimental): Salsalate, statin and omega-3-fatty acid combination therapy
  Interventions: Drug: Anti-inflammatory Combination Therapy

INTERVENTIONS:
Drug: Anti-inflammatory Combination Therapy — 1. salsalate: target dose 4 gm/day, administered in two divided doses of 2 gm in the morning and 2 gm in the evening
  2. fluvastatin: target dose 40 mg/day, administered in a single evening dose
  3. combined omega-3-fatty acid preparation of EPA and DHA; target dose EPA 2 gm/day and DHA 2 gm/day administered in a single evening dose
  Arms: Anti-inflammatory Combination Therapy
Drug: Placebo — Non-medication pills; To be taken in morning and evening intervals.
  Arms: Placebo

SUMMARY:
Despite current antipsychotic treatment, the majority of people with schizophrenia continue to exhibit persistent positive and negative symptoms and cognitive impairments. An alternative approach to the use of psychotropic agents for the treatment of persistent symptoms is the use of anti-inflammatory agents to reverse the pro-inflammatory state hypothesized to underlie the symptom and sign manifestations of the illness.

The investigators primary hypothesis is that add-on anti-inflammatory combination therapy will have significant beneficial effects on persistent positive symptoms and cognitive impairments.

The investigators secondary hypotheses are:

1. add-on anti-inflammatory combination therapy will be associated with improvements in depressive and negative symptoms and a reduction in pro-inflammatory cytokines
2. add-on anti-inflammatory combination therapy compared to placebo will not be associated with elevated adverse risk.

DETAILED DESCRIPTION:
Schizophrenia has been hypothesized to be due, in part, to disruptions of normal immune system and inflammatory responses to viral or bacterial infections or other stimuli of these systems. Epidemiological and clinical studies have provided extensive evidence that perinatal exposure to infection contributes to the etiology of schizophrenia. The recent reports of associations between markers of single nucleotide polymorphisms located within the major histocompatibility complex on chromosome 6p22.1 and schizophrenia provide further support for etiological hypotheses of immune system dysfunction in schizophrenia.

There are a large number of reports that suggest that people with schizophrenia have altered cytokine levels, with one or more studies reporting elevated levels of the pro-inflammatory cytokines: IL-1β, IL-6, IL-12, CRP, IFN-γ, and TNF-α; and reduced levels of the anti-inflammatory cytokine: IL-10. In this study we examine the use of combination anti-inflammatory therapy as an intervention in patients with schizophrenia. We will use

1. Salsalate, 4 gm/day. Salsalate is a potent inhibitor of nuclear transcription factor NF-κB activation. NF-κB is activated by pro-inflammatory cytokines;
2. Omega-3-fatty acids eicosapentaenoic (EPA; 2 gm/day) and docosahexaenoic (DHA; 2 gm/day). Omega-3-fatty acids exert their anti-inflammatory effects through their oxygenation into resolvins or protectins, which are potent anti-inflammatory agents;
3. Fluvastatin, 40 mgs/day. Fluvastatin is a lipid-lowering drugs, which acts through the inhibition of 3-hydroxy-3-methylglutaryl coenzyme A reductase (HMG-CoA). Fluvastatin may also exert anti-inflammatory effects independent of its lipid-lowering effects via a mechanism involving HMG-CoA inhibition and decreased NF-κB activation.

We have chosen to use combination therapy with three different classes of anti-inflammatory agents to address the potential benefit of this therapeutic approach for persistent positive symptoms and cognitive impairments. The three agents have unique anti-inflammatory mechanisms of action, which we believe offers the most robust evaluation of this therapeutic approach and maximizes the likelihood of eliciting pronounced therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants will meet DSM-IV-TR criteria for schizophrenia or schizoaffective disorder.
* Participants will be required to meet the following symptom criteria:

  1. BPRS total score of 45 or greater on the 18 item version (scale: 1-7) or a Clinical Global Impression (CGI) severity of illness item score of 4 (moderate) or greater.
  2. BPRS positive symptom item total score of 8 or greater and a score of 4 or more on at least one individual item.
* Participants will be clinically stable, be treated with the same antipsychotic for at least 60 days and a constant therapeutic dose for at least 30 days prior to study entry.
* Participants must be judged competent to participate in the informed consent process and provide voluntary informed consent

Exclusion Criteria:

* Participants who meet DSM-IV-TR criteria for alcohol or substance dependence (except nicotine) within the last 6 months or DSM-IV-TR criteria for alcohol or substance abuse (except nicotine) within the last month will be excluded
* Participants with a current infection or an organic brain disorder or medical condition, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol will be excluded.
* Participants with a history of: aspirin allergy, pre-existing tinnitus, tuberculosis, HIV, or hepatitis C; or autoimmune disease.
* Participants who are currently treated with a statin, warfarin, dipyridamole, or other anti-coagulants.
* Participant is currently treated with an omega-3-fatty acid preparation and cannot discontinue their use of the preparation for the duration of the study.
* Female participant who is sexually active and not using any form of birth control such as oral contraceptives or IUDs.
* Female participant who is pregnant or breastfeeding.
* Participant with current/active peptic ulcer disease or gastritis; anemia or thrombocytopenia (platelet count ≤120).
* Participant who is currently treated with a medication that can increase the risk of myopathy and rhabdomyolysis such as Fluconazole, Ketoconazole, Colchicine, Daptomycin, Erythromycin, or immunosuppressants that alter statin levels.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, MD, Principal Investigator — Maryland Psychiatric Research Center, University of Maryland School of Medicine; William T Carpenter, MD, Principal Investigator — Maryland Psychiatric Research Center, University of Maryland School of Medicine
Locations (1):
- Maryland Psychiatric Research Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Buchanan RW, Weiner E, Kelly DL, Gold JM, Chen S, Zaranski J, Blatt F, Wehring H, Carpenter WT. Anti-inflammatory Combination Therapy for the Treatment of Schizophrenia. J Clin Psychopharmacol. 2020 Sep/Oct;40(5):444-450. doi: 10.1097/JCP.0000000000001253. PMID 32796391

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Signed a consent form: 52 (50 unique subjects: 2 withdrew then later re-enrolled, not counted in analysis); Ineligible prior to Evaluation Phase: 1 subject (1=clinically unstable); Entered Evaluation Phase: 49 subjects; Withdrawn prior to randomization: 10 (8=Did not meet BPRS criteria; 1=Did not meet age criteria; 1=On an excluded medication)
Groups:
- Anti-inflammatory Combination Therapy: Salsalate, statin and omega-3-fatty acid combination therapy
  Anti-inflammatory Combination Therapy: a. salsalate: target dose 4 gm/day, administered in two divided doses of 2 gm in the morning and 2 gm in the evening b. fluvastatin: target dose 40 mg/day, administered in a single evening dose c. combined omega-3-fatty acid preparation of EPA and DHA; target dose EPA 2 gm/day and DHA 2 gm/day administered in a single evening dose
- Placebo: Placebo pills to be assigned using a permuted randomization system
  Anti-inflammatory Combination Therapy: a. salsalate: target dose 4 gm/day, administered in two divided doses of 2 gm in the morning and 2 gm in the evening b. fluvastatin: target dose 40 mg/day, administered in a single evening dose c. combined omega-3-fatty acid preparation of EPA and DHA; target dose EPA 2 gm/day and DHA 2 gm/day administered in a single evening dose
  Placebo: Non-medication pills; To be taken in morning and evening intervals.
Period: Overall Study
Arm/Group | Anti-inflammatory Combination Therapy | Placebo
Started | 19 | 20
Completed | 13 | 14
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-inflammatory Combination Therapy | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 18 | 18
  Not Hispanic or Latino | 19 | 1 | 20
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 10 | 9 | 19
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Persistent Positive Symptoms
Description: The Brief Psychiatric Rating Scale (BPRS) positive symptom items are: conceptual disorganization, hallucinatory behavior, unusual thought content, and suspiciousness. The total score is calculated by adding the scores for each item. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum score is 4 and the maximum score is 28. A higher score indicates a more severe positive symptom rating.
Time Frame: The BPRS will be administered at baseline and every two weeks throughout the double-blind phase of the study, for up to 12 weeks.
Population: Participants completing the BPRS assessment rating.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Anti-inflammatory Combination Therapy
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline Week 0 | 13 [12 to 16] | 14 [12 to 15]
  Treatment Week 2 | 14 [11 to 16] | 14 [11 to 18]
  Treatment Week 4 | 14 [10 to 16] | 15 [11 to 16]
  Treatment Week 6 | 14 [11 to 16] | 14 [12 to 15]
  Treatment Week 8 | 12 [10 to 16] | 14 [10 to 17]
  Treatment Week 10 | 14 [10 to 15] | 14 [10 to 16]
  Treatment Week 12 | 14 [10 to 15] | 12 [10 to 14]

2. Primary Outcome: Change in Neuropsychological Test Performance
Description: The MATRICS Consensus Cognitive Battery (MCCB) composite score by week ranging from -10-100 with a higher score indicating a better outcome.
Time Frame: The MCCB was administered at baseline and end-of-study (Week 12).
Population: Participants completing the MCCB testing.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Anti-inflammatory Combination Therapy
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline Week 0 | 25 [18.5 to 35] | 36 [24 to 48.5]
  Treatment Week 12 | 24 [20 to 29.2] | 26 [13.8 to 41.2]

3. Secondary Outcome: Change in Depressive Symptoms
Description: The Calgary Depression Scale (CDS) total score will be used to measure depressive symptoms. Total score calculated by adding scores for scales #1-#9. Each scale ranges from "0=Absent" to "3=Severe". The minimum total CDS score is 0 and the maximum total CDS score is 27. A higher score indicates a more severe depression rating.
Time Frame: The CDS was administered at baseline and every two weeks throughout the double-blind phase of the study, for up to 12 weeks.
Population: Participants completing the CDS assessment rating.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Anti-inflammatory Combination Therapy
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline Week 0 | 2 [0.5 to 3.5] | 0 [0 to 2]
  Treatment Week 2 | 2 [0 to 4] | 1 [0.75 to 2]
  Treatment Week 4 | 1 [0.25 to 3] | 1 [0 to 2.5]
  Treatment Week 6 | 2 [1 to 3] | 1 [0 to 3]
  Treatment Week 8 | 2 [1 to 2] | 1 [0 to 1]
  Treatment Week 10 | 2 [0 to 2] | 0 [0 to 1]
  Treatment Week 12 | 1 [0 to 2] | 0 [0 to 1.8]

4. Secondary Outcome: Change in Negative Symptoms
Description: The Scale for the Assessment of Negative Symptoms (SANS) total score, minus the global items, inappropriate affect, poverty of content of speech, and attention items, used to measure negative symptoms. Median SANS total score by treatment and week. SANS total score range = 0-85. Higher scores indicate more severe negative symptoms.
Time Frame: Baseline and every two weeks throughout the double-blind phase of the study, for up to 12 weeks.
Population: Participants completing the SANS rating assessment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Anti-inflammatory Combination Therapy
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline Week 0 | 27 [24 to 30] | 26 [19 to 34]
  Treatment Week 2 | 28 [23 to 33] | 24 [20 to 30]
  Treatment Week 4 | 32 [25 to 34] | 30 [20 to 34]
  Treatment Week 6 | 28 [21 to 34] | 27 [23 to 30]
  Treatment Week 8 | 30 [25 to 36] | 24 [19 to 34]
  Treatment Week 10 | 30 [24 to 33] | 30 [17 to 32]
  Treatment Week 12 | 28 [22 to 34] | 28 [19 to 32]

5. Secondary Outcome: Change in Pro-inflammatory Cytokines
Description: Data was only available on 2 of the 9 cytokines (i.e., IL-2 and IL-8) and C-Reactive Protein (CRP). The baseline values for the other cytokines in the panel were below the level of detection.
Time Frame: A cytokine profile will be collected at baseline and at week 12 (end-of-study).
Population: Participants who had a cytokine profile collected.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | Anti-inflammatory Combination Therapy
Number analyzed (Participants) | 19 | 19
pg/ml
  Baseline IL-2 levels | 59.16 (88.38) | 34.94 (77.01)
  End of study IL-2 levels | 88.4 (146.0) | 47.5 (86.0)
  Baseline IL-8 levels | 9.16 (5.59) | 8.35 (4.59)
  End of study IL-8 levels | 8.91 (7.24) | 19.78 (46.91)

6. Secondary Outcome: Change in C-Reactive Protein (CRP)
Description: as for outcome 5
Time Frame: A cytokine profile will be collected at baseline and at week 12 (end-of-study).
Population: Participants who had a cytokine profile collected.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Anti-inflammatory Combination Therapy
Number analyzed (Participants) | 19 | 19
ng/ml
  Baseline CRP levels | 38953 (27218) | 42950 (32468)
  End of study CRP levels | 38759 (21753) | 31849 (23176)

ADVERSE EVENTS:
Time Frame: 12-week Treatment Phase.
Description: Participants are systematically monitored for any increases on the Side Effects Checklist (SEC). An SEC AE includes any symptom/side effect rated with a score of 4 (severe) or for which there was a 2 point change in severity from baseline.
  Psychotic symptoms are also systematically monitored with the Brief Psychiatric Rating Scale (BPRS) rating. A BPRS AE includes an increase of 3 points or more relative to baseline or an increase from a score of 5 (moderately severe) to a 7 (very severe).
Arm/Group | Placebo | Anti-inflammatory Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/19
Other Adverse Events (participants affected / at risk) | 10/20 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Anti-inflammatory Combination Therapy (N=19)
Hospitalization (General disorders) | 0 (0) | 1 (1) — Hospitalized for acute febrile illness and Drug Rash with Eosinophilia and Systemic Symptoms (DRESS) syndrome. The fever and rash were judged to be possibly study drug related. The SAE resolved upon discontinuation of the study drugs.
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Hospitalization for worsening of clinical symptoms. The symptom exacerbation resolved with treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Anti-inflammatory Combination Therapy (N=19)
Eructation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (General disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Psychiatric symptom increase (Psychiatric disorders) | 4 (6) | 4 (8)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
High triglyceride levels (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abnormal EKG (Cardiac disorders) | 0 (0) | 1 (1)
Hypersalivation (General disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Fever (General disorders) | 0 (0) | 2 (2)
Upset stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Memory loss (General disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Myoclonus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (General disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Gait instability (General disorders) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dark urine (Renal and urinary disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Generalized pain (Nervous system disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT01514682/Prot_SAP_000.pdf